CLINICAL TRIAL: NCT02973971
Title: Pilot Study on Patients with Mild to Moderate Form of Alzheimer's Disease and Healthy Volunteers: Characterization of Intra-subject Variability and Chronobiological Variations of ADDIA Biomarkers.
Brief Title: ADDIA Chronobiological Study
Status: Completed | Type: Observational
Sponsor: Amoneta Diagnostics SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ST0055
Record Dates: First submitted 2016-11-15; First posted 2016-11-28 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
Keywords: Blood cell biomarkers, peripheral circulating biomarkers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy subjects
  Interventions: Other: volumeric MRI
- Alzheimer patients
  Interventions: Other: volumeric MRI

INTERVENTIONS:
Other: volumeric MRI

SUMMARY:
The present single center clinical chronobiological study on 24 subjects (12 patients with mild to moderate form of Alzheimer's disease and 12 Healthy subjects) aims at characterizing the ADDIA biomarkers: a) blood cell-based biomarkers measured by flow cytometry using proprietary probes specific of two targeted biomarkers, beta-Amyloid (Aβ) peptide and a kinase, and b) circulating biomarkers in peripheral body fluids. The biomarkers will be analyzed on samples taken at different time points of the day, including under fasting and non-fasting conditions and at two periods: day 1 and day 14.

ELIGIBILITY:
Inclusion Criteria for Alzheimer patient group:

* Signed Informed Consent.
* Male or female subject, between 55 and 85 years inclusive.
* Specific clinical phenotype of AD: Presence of an early and significant episodic memory impairment (isolated or associated with other cognitive or behavioural changes that are suggestive of a dementia syndrome) that includes the following:

  * Gradual and progressive change in memory function reported by patient or informant over more than 6 months.
  * Objective evidence of an amnesic syndrome of hippocampal type, based on significantly impaired performance on an episodic memory test with established specificity for mild to moderate AD.
* Cognitive tests including MMSE score 12 ≤ MMSE ≤ 25 for mild to moderate AD (measured in the last 3 months), b) Scores of other tests routinely practiced at the hospital for measurement of memory and cognition shall be compatible with mild to moderate AD.
* Neuroimaging compatible with a diagnosis of mild to moderate AD.
* Cerebrospinal fluid (CSF) biomarkers showing at least 2 positive levels out of the 3 biomarkers: CSF Aβ1-42 and tau (Phosphorylated-Tau and/or Total-Tau). CSF collection and data being only retrospective.

Inclusion Criteria for healthy controls:

* Signed Informed Consent.
* Male or female subject, between 55 and 85 years inclusive.
* Normal clinical and cognitive scores as measured using standard neuropsychological tests.
* Normal scores in other neuropsychological tests routinely practiced at the hospital for measurement of memory and cognition.
* No abnormal neuroimaging findings in at least structural MRI.

Exclusion Criteria:

* Any subject who did not sign the informed consent form.
* Any chronic neurodegenerative disease (vascular dementia, Parkinson's disease, Creutzfeldt Jacob, Huntington's disease, etc.), acute neurodegenerative disease (stroke), history or presence of clinically relevant psychiatric history (schizophrenia, psychosis), some chronic inflammatory diseases that impact blood cells (e.g. anemia of inflammation and chronic disease) and some cancers (that impact blood cells: e.g. leukemia), major sensory deficits that could interfere with cognitive assessment (visual and auditory), epilepsy.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Neutropenia (Neutrophils < 1500/mm3).
* Thrombocytopenia (platelets: < 100,000/mm3, rule out EDTA-induced pseudothrombocytopenia).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 12 patients with mild to moderate form of Alzheimer's disease 55 to 85 years-old.
  * 12 healthy volunteers (HV), 55 to 85 years-old.
  * Total expected completed subjects: 24.
  * Stratification by gender: 6 males and 6 females, age-matched healthy subjects and 6 males and 6 females, age-matched Alzheimer patients.
  * Mean age similar in both groups
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Blood cell biomarker level | Two weeks
  To characterize the targeted blood cell biomarkers by assessing the effects of effect of meal, age and gender on biomarkers and changes in biomarker expression levels over two periods (day 1, day 15).

SECONDARY OUTCOMES:
Circulating biomarker level | two weeks
  To characterize the circulating biomarkers by assessing the effects of effect of meal, age and gender on biomarkers and changes in biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Blanc, MD, Principal Investigator — Hôpitaux Strasbourg; Catherine Mutter, MD, Principal Investigator — Hôpitaux Strasbourg
Locations (1):
- Hopitaux Universitaires de Strasbourg, Strasbourg, Alsace, France

IPD SHARING:
Plan to Share IPD: No